CLINICAL TRIAL: NCT04487977
Title: International Survey on Airway Management in COVID-19 Patients (ISAM-COVID)
Brief Title: Survey on COVID-19 Airway Management
Acronym: ISAM-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spanish Society of Anesthesia and Critical Care (SEDAR) (Other)
Collaborators: Confederation of Latin American Societies of Anaesthesiology (CLASA) (Unknown)
Responsible Party: Principal Investigator, Dr. Manuel Granell Gil, Professor, Spanish Society of Anesthesia and Critical Care (SEDAR)
Other Study IDs: ISAM-COVID
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Airway Management
Keywords: airway; COVID-19; critical care; anesthesia; airway management
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Surveyed professionals
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Answering a survey on airway management in COVID-19 patients

SUMMARY:
The objectives of this study are to analyze the best device for intubation in patients infected by SARS-CoV2 virus during COVID-19 pandemics and to review the optimal methods for airway management in such patients for elective surgery and in the Critical Care environment. Also, the safest methods for airway management in thoracic surgery will be analyzed.

This study has a descriptive design with no hypothesis contrast, and it will explore the current picture in airway management in Spain. It is a multicentric international study, for all the centers where intubations of tracheostomies have been performed in patients diagnosed with SARS-CoV2 with positive PCR, either in the Critical Care setting or the operating room.

A survey will be distributed among professionals who have been involved in airway management in COVID-19 patients in the following specialties: Anesthesiology and Critical Care Medicine, Emergency Medicine, Prehospital Medicine, Cardiology and Pulmonology.

The study started on april 2020 after receiving approval from the Ethics Committee (General University Hospital of Valencia) COVID-19 infection causes respiratory failure needing ventilatory support, which required endotracheal intubation or tracheostomy. This situation poses a significant risk of transmission due to its usual urgent nature, and it often happens in the context of respiratory claudication. For this reason, studying the safest and useful methods for airway management in this kind of patients, using data based on the clinical experience, may be of great interest in the future.

Statistical analysis will be performed using Statistical Software R, . Technical characteristics will be described using frequencies and percentages for categorical variables, and means and standard deviations or medians and interquartile ranges for continuous variables, depending on normality tests. Base characteristics, center and years of experience will be compared.

A sample size calculation is not necessary, since it is an explorative and voluntary study, trying to establish which are the regular routines in airway management in COVID-19 patients in Spain and Latin America.

DETAILED DESCRIPTION:
1. Justification There are no studies about safety and effectiveness of different airway management procedures in COVID-19 patients in Spain or Latin America.

   Due to the emergent nature of this disease, there are very few solid and universal publications about safety or validated protocols in SARS-CoV-2 disease airway management.

   In the last months, and following the clinical experience coming from China and Italy, we have been able to see how SARS-CoV-2 virus has caused severe morbidity or death in thousands of patients. In this line, and considering the high transmission rate of this disease, we observe how professionals from these countries have performed airway management to provide proper ventilation and oxygenation, in either potentially critically ill patients or in a surgical context. Their experience has allowed other countries to develop specific protocols, and to quickly adapt them to the updates that keep happening daily.

   For this reason, we want to explore the Spanish and Latin American experience in airway management. It is important to draw conclusions not only from the preparations and technical approaches, but also the information stemming from the context in which the procedure is performed, the stress derived from the risk of transmission and the personal protective equipment, as well as the particular difficulties they add to the technique.
2. Hypothesis: Since it is a descriptive study, there is no formal hypothesis in this work.

   Objectives
3. Objectives:

   3.1. Main objective: To analyze the preferred device for intubation in patients infected by SARS-CoV2 virus during COVID-19 pandemics using a survey addressed to health care professionals experienced in assistance to COVID-19 patients. The preferred device will be rated using an ordinal scoring scale and it will be presented as the device with the highest score.

   3.2. Secondary objectives: To assess the preferred methods for airway management in COVID-19 patients in a Critical Care setting or undergoing urgent or elective surgery.
4. Design: Descriptive design with no hypothesis contrast, exploring the current panorama in airway management in Spain and Latin America.
5. Ambit: Multicenter and international for Spain and Latin America, for all the health care centers where intubations or tracheostomies have been performed in COVID-19 patients with a positive PCR, either in the Critical Care setting or in the operating room.
6. Study population: The study population will consist of all the health care professionals who have been or are currently involved in airway management in COVID-19 positive patients, from the following medical specialties: Anesthesiology and Critical Care Medicine, Emergency Medicine, Pre-Hospital Medicine, Cardiology, Pulmonology.
7. Variables:

   7.1. Main variable: Optimal device: Which is the best rated device for endotracheal intubation in COVID-19 patients.

   7.2. Secondary variables:
   * Context in which the professional has experience when intubation COVID-19 patient: 1. Critical Context (Emergency Department, Critical Care Unit), 2. Emergent Surgery, 3. Elective Surgery.
   * Professional opinion about the usefulness of different systems for reducing aerosol production or diffusion (from 1 to 6, where 1 is the least useful and 6 is the most useful): 1. Methacrylate box with accesses for the arms, 2. Face mask tight seal, 3. Negative pressure system in the intubation area, 4. Avoidance of hand ventilation, 5. Rapid sequence intubation, 6. Sellick maneuver, 7. Other.
   * Professional opinion about the importance of the different drawbacks of video laryngoscopes (from 1 to 6, where 1 is the most important and 6 is the least important): 1. Reflections on the screen, 2. Difficulty to introduce the blade in the mouth, 3. Proximity to the patient's airway, 4. Difficulty to insert the tube through the vocal cords, 5. Lack of experience with the specific video laryngoscope used, 6. Preference for direct laryngoscopy due to higher experience and confidence with it.
   * Type of blade most often used by use: 1. Reusable, 2. Disposable.
   * Type of blade most often used by channel: 1. With channel, 2. Without channel.
   * Type of blade most often used by curvature: 1. Regular curve, 2. Hyper Curved.
   * Type of video laryngoscope screen: 1. Integrated with the main device, 2. Away from the device.
   * Type of aid device (from 1 to 6, where 1 is the least useful and 6 is the most useful): 1. Frova introducer, 2. Eschman introducer, 3. Flexible introducer inside the tube, 4. Flexible endoscope, 5. VAMA, 6. Other.
   * Preferred method for intubation in the foreseen difficult airway situation (from 1 to 6, where 1 is the most preferred and 6 is the least preferred): 1. Fiberoptic intubation, 2. Intubation with video laryngoscope, 3. Direct laryngoscopy, 4. McCoy laryngoscope, 5. Intubation through a laryngeal mask, 6. Tracheostomy.
   * Preferred method for intubation in the unforeseen difficult airway situation (from 1 to 6, where 1 is the least preferred and 6 is the most preferred):1. Fiberoptic intubation, 2. Intubation with video laryngoscope, 3. Direct laryngoscopy, 4. McCoy laryngoscope, 5. Intubation through a laryngeal mask, 6. Tracheostomy.
   * Preferred strategies upon surgical conclusion in COVID-19 patients (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. To extubate all patients in the Critical Care Unit, 2. To extubate all patients in the operating room, 3. To extubate only stable patients in the operating room, if postoperative ventilation os not expected, 4. Other.
   * Preferred procedures in intubated COVID-19 patients who need a tracheostomy (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. Open conventional tracheostomy, 2. Percutaneous tracheostomy, 3. Fiberoptic guidance to conduct location and opening of the trachea, 4. Apnea or ventilator stand-by for as long as possible.
   * Professional rating of different assertions about techniques and equipment to intubate COVID-19 patients (from 1 to 6, where 1 is the lowest validity and 6 is the highest validity): 1. It is concerning to use reusable material with the possibility of contamination, 2. It is concerning to move intubation equipment from COVID-19 to non-COVID-19 areas, 3. Swiftly intubating critical or severely deteriorated COVID-19 patients is related to a higher risk of transmission, 4. Airway management maneuvers with personal protective equipment are more difficult and uncomfortable.

   Specific variables in the thoracic surgery context, to be answered only by professionals working with such patients:
   * Experience in thoracic anesthesia: 1. Over 10 years, 2. From 5 to 10 years, 3. Under 5 years, 4. No experience.
   * Preferred method to perform lung isolation in COVID-19 patients (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. Conventional double lumen tubes and flexible endoscope, 2. Double lumen tubes with attached camera, 3. Bronchial blocker, endotracheal tube and flexible endoscope, 4. Bronchial blocker and endotracheal tube with attached camera (Viva Sight ®), 5. Univent ® tube and flexible endoscope, 6. Other.
   * Preferred video laryngoscope for double lumen tube insertion in COVID-19 patients with a difficult airway (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. C-MAC ®, 2. King Vision ®, 3. McGrath ®, 3. GlideScope ®, 4. Airtraq ®, 5. Other.
   * Preferred bronchial blocker for COVID-19 patients (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. Arndt, 2. Cohen, 3. Univent ® tube, 4. EZ Blocker ®, 5. Fogarty catheter, 6. Other)
   * Preferred position for the antiviral /antibacterial filter (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. Expiratory branch, 2. Inspiratory branch, 3. Y bifurcation, 4. Proximal end of the endobronchial lumen of the double lumen tube, leading to the non ventilated lung to be collapsed, 5. Proximal end of the bronchial blocker, if it is used.
   * Usefulness of the closed and regulable aspiration system for the non ventilated lung: 1. Yes, 2. No.
   * Preferred strategies upon surgical conclusion in COVID-19 patients (from 1 to 6, where 1 is the least preferred and 6 is the most preferred): 1. To extubate all patients in the Critical Care Unit, 2. To extubate all patients in the operating room, 3. To extubate only stable patients in the operating room, if postoperative ventilation os not expected, 4. To exchange the double lumen tube for an endotracheal tube and extubation in the post anesthesia unit, 5. To withdraw the double lumen tube to the trachea for subsequent extubation in the post anesthesia unit, 6. To remove the bronchial blocker and leave the endotracheal tube for subsequent extubation in the post anesthesia unit, 7. To remove the bronchial blocker from the Univent ® tube and subsequent extubation in the post anesthesia unit, 8. Other.
   * Number of intubations performed in COVID-19 patients.
   * Personal SARS-CoV-2 infection: 1. Yes, 2. No.
8. Information sources: Variables will be obtained from a voluntary survey accessible from the Internet, created with Microsoft Forms ®. Microsoft Forms ® is a digital platform with a free access plan which allows quick and development of digital surveys with no need for programming. It also includes a set of tools to distribute and gather the results from the questionnaires. The survey is accessed from a link sent via e-mail or other digital distribution methods to the potential participants.
9. Interventions and procedures: There is no need for interventions on patients or their clinical records. A single intervention will take place on the participants in the moment of sending the survey. This only contact will provide all the aforementioned variables.
10. Sample size calculation: There is no need for sample size calculation, since the study is explorative and voluntary, trying to assess clinical routines in airway management.
11. Statistical plan: Statistical analysis will be performed using Statistical Software R, . Technical characteristics will be described using frequencies and percentages for categorical variables, and means and standard deviations or medians and interquartile ranges for continuous variables, depending on normality tests. Base characteristics, center and years of experience will be compared. Proper figures will be presented to represent the results about which are the most used techniques and devices, as well as the most important features of every procedure.
12. Ethical considerations:

12.1. General considerations: The study is to be conducted according to this protocol, Helsinki Ethical Principles Declaration and currently existing directives.

12.2. Informed consent: An informed consent form is not necessary, since the survey will be completed by professionals who provided care to the patients in a retrospective manner, with no diagnostic or therapeutic interventions. Besides, since it is a retrospective study with anonymous data, there is no possibility to ask for an informed consent to the patients. For these reasons, an exemption for informed consent was requested and accepted by the Ethics Committee.

12.3. Data protection: Data from the participants will be managed according to existing spanish and european laws (Spanish Law 3/2018 on Personal Data Protection and Digital Rights Warranty, and EU Regulation UE 2016/679). Gathered data for the study will be identified with a code, and the information will not include identificatory details of the participants, thus not being able to reveal their identities. Names of patients will not be collected or presented in any publication or communication of the study results.

ELIGIBILITY:
Inclusion Criteria: Professionals belonging to medical specialties involved in airway management who have performed intubation and/or tracheostomy maneuvers in COVID-19 patients during current pandemics.

Exclusion Criteria:

* Professionals not belonging to medical specialties involved in airway management or with no experience in intubation/tracheostomy maneuvers.
* Those not willing to answer the survey.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Professionals belonging to medical specialties involved in airway management who have performed intubation and/or tracheostomy maneuvers in COVID-19 patients during current pandemics.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Preferred device | During COVID-19 pandemics in each country, since the release of the survey until its closure, approximately 4 months
  Preferred device for intubation in COVID-19 patients infected by SARS-CoV2

CONTACTS AND LOCATIONS:
Locations (1):
- Consorcio Hospital General Universitario de Valencia, Valencia, Spain